CLINICAL TRIAL: NCT06228222
Title: Predictors of Remission and Renal Outcomes in Lupus Nephritis in Assuit University Hospitals.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Athanassios Faraj Manassa, student, Assiut University
Other Study IDs: Predictors of remission in LN.
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus
Keywords: lupus nephritis; systemic lupus erythematosus; predictors of outcomes
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: patients with lupus nephritis who will be admitted to Rheumatology and Nephrology Units, Internal Medicine Department, Assuit university hospitals, Egypt. (classified according to the 1997 American College of Rheumatology or Systemic Lupus Collaborating Clinics criteria) with biopsyproven LN (classified according to The revised ISN/RPS 2018mhistopathological classification system).
  Interventions: Procedure: renal biopsy

INTERVENTIONS:
Procedure: renal biopsy — Renal biopsy will be performed for all patients fulfilling the American College of Rheumatology (ACR) criteria to confirm the diagnosis of lupus nephritis (LN) and to classify the glomerular disease by "the revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2018 histopathological classification system"

SUMMARY:
the goal of this opservetional study is to identify predictors of remission and renal outcomes in SLE patients affected with Lupus nephritis. the main question it aims to answer is:

*What are the clinical, histological and chemical parameters that connected to undesirable renal prognosis in LN?

All patients will be subjected to the following:

Complete through history taking, clinical examination disease activity will be assessed by SLEDAI. The Laboratory investigations and renal biopsy.

DETAILED DESCRIPTION:
Systemic lupus erythematosus is a chronic, multisystemic, inflammatory, autoimmune disorder characterized by the formation of autoantibodies directed against self-antigen and immune complex resulting in a wide range of clinical manifestations and target organs (kidney, lungs) damage with unpredictable flares and remissions that eventually lead to permanent injury Lupus nephritis( LN ) is one of the most severe complications in SLE, affecting 35 %- 60 % of the individuals depending on ethnicity, sex, age at the onset of the disease, Course of SLE disease, hereditary factors and nephron cargo and renal toxicity(drug - induced toxicity for example), add to long - term damage of the renal function. LN flares constitute a significant cause of nephron loss, contributing to renal function loss. Recent therapies for LN are not sufficiently effective in preventing or inducing recovery. flares and not all patients show sufficient treatment actions. In fact, fewer than 30 % achieve full recovery within 6 months of treatment. Up to 20 % of patients in recent decades have been affected by LN will eventually develop end - stage renal disease within the first decade of their disease's progression. For this reason, Prediction of the long - term renal outcomes at early stages of the disease is of critical importance. Therefore, many studies have sought to identify early clinical characteristics, lab tests and chemical processes that are connected to undesirable renal prognosis, in order to optimize the monitoring and interventions in these patients. The goals of management of individuals with LN may be divided into short - term ( reduction of flares ) and long - term targets( prevention of renal function impairment ). Currently conducted studies in the field focuses on identifying of clinical, histological and chemical signs of action, damage, treatment response and renal function outcome

All patients will be subjected to the following:

Complete through history taking, clinical examination disease activity will be assessed by SLEDAI. The Laboratory investigations, reported at the time of renal biopsy and after 1, 3, 6 months of treatment:

1. complete blood count,
2. serum creatinine (SCr)
3. SLEDAI
4. serum albumin
5. C-reactive protein
6. urine analysis
7. 24-hour urinary protein excretion
8. glomerular filtration rate ( eGFR)
9. C3 and C4 levels and autoantibody profile, including ANA and anti-dsDNA antibodies,
10. Renal biopsy:

Renal biopsy will be performed for all patients fulfilling the American College of Rheumatology (ACR) criteria to confirm the diagnosis of lupus nephritis (LN) and to classify the glomerular disease by "the revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2018 histopathological classification system" Also, LN class and activity and chronicity scores will be recorded. Patients will be reviewed at one month, three months, and six months for clinical assessment, renal function assessment (SCr and eGFR), assessment of proteinuria, and monitoring response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and SLE patients with biopsy-proven LN.

Exclusion Criteria:

* Severe physical disability, patients with uncontrolled hypertension, diabetes mellitus, or severe ischemic heart diseases, patients with mental illness, patients with overlap syndrome, and refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study to be conducted on SLE patients with lupus nephritis who will be admitted to Rheumatology and Nephrology Units, Internal Medicine Department, Assuit university hospitals, Egypt. the SLE patients (classified according to the 1997 American College of Rheumatology or Systemic Lupus Collaborating Clinics criteria) with biopsyproven LN (classified according to The revised ISN/RPS 2018 histopathological classification system).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission | 25 jan 2024 to 1 oct 2025.
  is defiened as albumin 35 g/l, urinary protein creatinine ratio (UPCR)<0.3g/g, a normal range of SCr or at a level increasing no more than 15% from baseline, and without lupus flares
partial remission | 25 jan 2024 to 1 oct 2025.
  is defined as albumin 30 g/l, a proteinuria > 0.3 but < 3.5 g per 24 hours or decrease 50% from baseline, a normal range of SCr or at a level increasing no more than 25% from the baseline and without lupus flares.
no remission no remission | 25 jan 2024 to 1 oct 2025.
  is defined as not meeting the response criteria.

REFERENCES:
- [Background] Parodis I, Tamirou F, Houssiau FA. Prediction of prognosis and renal outcome in lupus nephritis. Lupus Sci Med. 2020 Feb 18;7(1):e000389. doi: 10.1136/lupus-2020-000389. eCollection 2020. PMID 32153796
- [Background] McDonald S, Yiu S, Su L, Gordon C, Truman M, Lisk L, Solomons N, Bruce IN; MASTERPLANS Consortium. Predictors of treatment response in a lupus nephritis population: lessons from the Aspreva Lupus Management Study (ALMS) trial. Lupus Sci Med. 2022 May;9(1):e000584. doi: 10.1136/lupus-2021-000584. PMID 35640982
- [Background] Herath N, Ratnatunga N, Weerakoon K, Wazil A, Nanayakkara N. Clinicopathological findings, treatment response and predictors of long-term outcome in a cohort of lupus nephritis patients managed according to the Euro-lupus regime: a retrospective analysis in Sri Lanka. BMC Res Notes. 2017 Feb 2;10(1):80. doi: 10.1186/s13104-017-2402-6. PMID 28148285
- [Background] Yadav S, Balakrishnan C, Kothari J. Long-term outcome and predictors of long-term outcome in patients with lupus nephritis managed at a tertiary hospital in Mumbai. Lupus. 2022 Sep;31(10):1191-1201. doi: 10.1177/09612033221106607. Epub 2022 Jun 4. PMID 35658736